CLINICAL TRIAL: NCT03892200
Title: Adapting an Evidence-Based Program That Improves Oral Hygiene and Health for Assisted Living Residents With Dementia
Brief Title: Oral Hygiene in Assisted Living
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-2795; R01AG061966 (NIH)
Record Dates: First submitted 2019-03-22; First posted 2019-03-27 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-03

CONDITIONS: Aging; Long-Term Care
Keywords: Mouth Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aim2 - Daily Mouth Care (Experimental): The intervention being tested is a standardized educational and skill-building program for use in assisted living communities, which highlights that mouth care is infection control (e.g., can reduce pneumonia); includes techniques and products to clean and protect the teeth, tongue, gums, and dentures (e.g., the jiggle-sweep approach to remove plaque, use of an interdental brush instead of floss); provides strategies for care provision in special situations (e.g., broken teeth); and includes a toolkit of dementia-sensitive approaches for people who are resistant (e.g., refuse to open the mouth). It also includes information about potential dental emergencies and issues that merit assessment.
  For Aim2 the intervention training is delivered by a research dental hygienist.
  Interventions: Behavioral: Aim2 - Daily Mouth Care
- Aim2 - Standard Mouth Care (No Intervention): Assisted living communities will continue to provide standard mouth care to all residents. Assisted living staff will not receive training or supplies in the control condition.
- Aim3 - Daily Mouth Care (Experimental): The intervention being tested is a standardized educational and skill-building program for use in assisted living communities, which highlights that mouth care is infection control (e.g., can reduce pneumonia); includes techniques and products to clean and protect the teeth, tongue, gums, and dentures (e.g., the jiggle-sweep approach to remove plaque, use of an interdental brush instead of floss); provides strategies for care provision in special situations (e.g., broken teeth); and includes a toolkit of dementia-sensitive approaches for people who are resistant (e.g., refuse to open the mouth). It also includes information about potential dental emergencies and issues that merit assessment.
  For Aim3 the intervention training is delivered by state public health dental hygienists.
  Interventions: Behavioral: Aim3 - Daily Mouth Care
- Aim3 - Standard Mouth Care (No Intervention): Assisted living communities will continue to provide standard mouth care to all residents. Assisted living staff will not receive training or supplies in the control condition.

INTERVENTIONS:
Behavioral: Aim2 - Daily Mouth Care — Nursing assistants will be trained to provide daily mouth care to all residents in nursing homes. Mouth care supplies will also be provided to intervention assisted living communities.
  For Aim2 the intervention training is delivered by a research dental hygienist.
  Arms: Aim2 - Daily Mouth Care
Behavioral: Aim3 - Daily Mouth Care — Nursing assistants will be trained to provide daily mouth care to all residents in nursing homes. Mouth care supplies will also be provided to intervention assisted living communities.
  For Aim3 the intervention training is delivered by state public health dental hygienists.
  Arms: Aim3 - Daily Mouth Care

SUMMARY:
This project will modify a program that reduces pneumonia among nursing home residents with dementia, so that it is appropriate for assisted living residents with dementia. The program provides daily mouth care to reduce bacteria in the mouth that lead to aspiration pneumonia. The project will develop methods that can be taught to assisted living providers by community dental hygienists, and that are ready for evaluation in a pragmatic trial of AL residents with dementia and the staff who provide their care.

DETAILED DESCRIPTION:
It could be said that many dementia care and caregiver support interventions are too limited, focusing solely on psychosocial and behavioral concerns. These issues are important, but so too is the physical health of people with dementia -- especially because they are living longer and require more support with health care and activities of daily living. Just imagine the benefit of a physical health care intervention provided daily.

Case in point: tooth brushing, flossing, and gum and denture care. Many people with dementia resist mouth care - almost 90% in nursing homes, in fact. As a result, only 16% have their teeth brushed regularly, putting them at risk for aspiration pneumonia when they inhale bacteria from their teeth, tongue, and gums. In 2013, the research team submitting this proposal developed one of the two existing dementia-focused mouth care programs for nursing homes -- Mouth Care Without a Battle (MCWB) -- which already has become a standard of nursing home care. MCWB changes caregivers' attitudes and behavior, improves oral health, and in a cluster randomized trial, MCWB provided by nursing assistants reduced pneumonia incidence by 32 percent.

The next frontier is to extend MCWB to assisted living (AL), the primary long-term residential care provider for persons with dementia. There are 30,200 AL communities across the country; 90% of their 835,200 residents have cognitive impairment and 42% have moderate or severe dementia (and on average, five untreated oral health conditions), meaning MCWB has the potential to improve the health and quality of life of more than 350,000 AL residents with dementia annually.

There is a unique and timely opportunity to transform MCWB so it is optimally suitable for AL, given the North Carolina Department of Health and Human Services (DHHS) Special Care Dentistry Program offer of partnership. Consequently, the investigators propose this nested cohort cluster randomized trial that will apply the NIH Stage Model and principles of the Science of Behavior Change (SOBC) to lay the groundwork for a pragmatic trial and real-world implementation of MCWB for AL residents with dementia and their caregivers.

The aims of the proposed project are to refine MCWB (NIH Stage I/Aim 1), and examine research efficacy (NIH Stage II/Aim 2) and real-world efficacy (NIH Stage III/Aim 3), focusing on structural, social, and interpersonal mechanisms as the SOBC target. Aims 2 and 3 will use separate samples of AL communities (24 for Aim 2 and 28 for Aim 3) across the state's ten regions. Within each region, one-half of AL communities will be randomized to treatment (MCWB) and one-half to control, and the oral hygiene of up to 360 residents with dementia will be assessed through eight months. For Aim 3 there will be up to 233 residents assessed for four months. In Aim 2, a research dental hygienist will train AL staff on MCWB and provide ongoing support; in Aim 3, this responsibility will be transferred to community public health dental hygienists working with the DHHS. Family members (one per resident, up to 360 for Aim 2 and up to 233 for Aim 3) will also be interviewed about the resident. Assisted Living staff will also be interviewed at each baseline and follow-up visit (up to 360 for Aim 2 and up to 360 for Aim 3).

Aim 1. Refine MCWB for implementation in assisted living (AL) communities.

1. Identify stakeholder perspectives. Interview (1) the administrator, health care supervisor, and a personal care aide (PCA) from 20 AL communities across North Carolina who have already been trained in MCWB by community-based public health dental hygienists from the DHHS Special Care Dentistry Program, and (2) the dental hygienists who provided that training, to learn attitudes regarding MCWB as developed for nursing homes, the extent to which care has changed, and recommended modifications to MCWB for AL.
2. Create a one-hour MCWB training video (web and digital versatile disc format) targeted to AL. Modifications include videorecording AL staff providing mouth care to residents with dementia, and interviews with residents and families; AL administrators, supervisors and PCAs; and dental hygienists.

Aim 2. Evaluate research efficacy of the MCWB program, with training and support provided by an experienced research dental hygienist.

1. Evaluate MCWB in terms of (1) the reach of the intervention; (2) effects on mediators/targets of change at the organizational and individual level; (3) resident outcomes (oral hygiene, pneumonia, hospitalizations); (4) associations between change at the organizational and individual level and outcomes, and also associations with characteristics of the AL community and staff; and (5) attitudes, barriers, and facilitators.
2. Develop a coaching manual for community hygienists to provide training and support to AL staff, reflecting lessons-learned from analyses.

Aim 3. Evaluate real-world efficacy of the MCWB program, transferring responsibility for training and support to community public health dental hygienists, thereby testing efficacy of a nationally generalizable model.

1. Assess dental hygienists' (up to N=24) self-efficacy to provide training and support at baseline and 4 months.
2. Evaluate MCWB as per Aim 2a, including examining associations with characteristics of the hygienists.
3. Compare implementation and effectiveness outcomes between research and real-world efficacy.
4. Refine the coaching manual for community dental hygienists to provide training and coaching, reflecting lessons-learned from analyses.

By the conclusion of this project, MCWB will be ready for evaluation in a pragmatic trial of AL residents with dementia and the staff who provide their care.

Note that the CT.gov record includes only the assisted living residents enrolled in the clinical trial, not secondary participants (staff, hygienists).

ELIGIBILITY:
RESIDENTS

Inclusion Criteria:

* Are 18 years of age or older
* Have teeth or have and use a denture
* Have a diagnosis of dementia

Exclusion Criteria:

* Requires antibiotic prophylaxis prior to oral hygiene examination
* Currently on hospice or tube-feeding
* Expected to die or be discharged in the next six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-03-13 (Actual)

PRIMARY OUTCOMES:
Aim2 - Plaque Index Score for Long-Term Care (PI-LTC) - Baseline | Baseline Visit
  The Plaque Index for Long-Term Care (PI-LTC) is a modification of the Simplified Oral Hygiene Index. It is derived by separately scoring the buccal and lingual surfaces of six sextants in the mouth (left, front, and right regions of the upper and lower jaw), resulting in 12 separate observations for residents with a full set of teeth; sextants not containing teeth do not receive a score. Within each sextant, the tooth surface with the worst plaque is scratched using an explorer and assigned a score (0=no plaque or stain present; 1=soft plaque covering not more than one third of the tooth surface or presence of extrinsic stains without other plaque regardless of surface area covered; 2=soft plaque covering between one third and two thirds of the tooth surface; or 3=soft plaque covering more than two thirds of the exposed tooth surface). PI-LTC scores range from 0-3 and are the average sextant score. Lower scores are better.
Aim2 - Plaque Index Score for Long-Term Care (PI-LTC) - 4 Months | 4 Months Follow-up Visit
  The Plaque Index for Long-Term Care (PI-LTC) is a modification of the Simplified Oral Hygiene Index. It is derived by separately scoring the buccal and lingual surfaces of six sextants in the mouth (left, front, and right regions of the upper and lower jaw), resulting in 12 separate observations for residents with a full set of teeth; sextants not containing teeth do not receive a score. Within each sextant, the tooth surface with the worst plaque is scratched using an explorer and assigned a score (0=no plaque or stain present; 1=soft plaque covering not more than one third of the tooth surface or presence of extrinsic stains without other plaque regardless of surface area covered; 2=soft plaque covering between one third and two thirds of the tooth surface; or 3=soft plaque covering more than two thirds of the exposed tooth surface). PI-LTC scores range from 0-3 and are the average sextant score. Lower scores are better.
Aim2 - Change in Plaque Index Score for Long-Term Care (PI-LTC) - 4 Months | Change from Baseline to 4 months
  The Plaque Index for Long-Term Care (PI-LTC) is a modification of the Simplified Oral Hygiene Index. It is derived by separately scoring the buccal and lingual surfaces of six sextants in the mouth (left, front, and right regions of the upper and lower jaw), resulting in 12 separate observations for residents with a full set of teeth; sextants not containing teeth do not receive a score. Within each sextant, the tooth surface with the worst plaque is scratched using an explorer and assigned a score (0=no plaque or stain present; 1=soft plaque covering not more than one third of the tooth surface or presence of extrinsic stains without other plaque regardless of surface area covered; 2=soft plaque covering between one third and two thirds of the tooth surface; or 3=soft plaque covering more than two thirds of the exposed tooth surface). PI-LTC scores range from 0-3 and are the average sextant score. Lower scores are better.
Aim2 - Gingival Index Score for Long-Term Care (GI-LTC) - Baseline | Baseline Visit
  The Gingival Index for Long-Term Care (GI-LTC) is a modification of the Gingival Index. Within each sextant, the most inflamed gingival surface is identified, swept using an explorer, and assigned a score (0=no inflammation; 1=mild inflammation, slight change in color, little change in texture; 2=moderate inflammation, glazing, redness, edema, and/or hypertrophy; or 3=severe inflammation, marked redness, edema and/or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration). Overall GI-LTC scores range from 0-3 and are the average sextant score. Buccal and lingual surfaces scores also are calculated. Lower scores are better.
Aim2 - Gingival Index Score for Long-Term Care (GI-LTC) - 4 Months | 4 Months Follow-up Visit
  The Gingival Index for Long-Term Care (GI-LTC) is a modification of the Gingival Index. Within each sextant, the most inflamed gingival surface is identified, swept using an explorer, and assigned a score (0=no inflammation; 1=mild inflammation, slight change in color, little change in texture; 2=moderate inflammation, glazing, redness, edema, and/or hypertrophy; or 3=severe inflammation, marked redness, edema and/or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration). Overall GI-LTC scores range from 0-3 and are the average sextant score. Buccal and lingual surfaces scores also are calculated. Lower scores are better.
Aim2 - Change in Gingival Index Score for Long-Term Care (GI-LTC) - 4 Months | Change from Baseline to 4 Months
  The Gingival Index for Long-Term Care (GI-LTC) is a modification of the Gingival Index. Within each sextant, the most inflamed gingival surface is identified, swept using an explorer, and assigned a score (0=no inflammation; 1=mild inflammation, slight change in color, little change in texture; 2=moderate inflammation, glazing, redness, edema, and/or hypertrophy; or 3=severe inflammation, marked redness, edema and/or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration). Overall GI-LTC scores range from 0-3 and are the average sextant score. Buccal and lingual surfaces scores also are calculated. Lower scores are better.
Aim2 - Denture Plaque Index Score (DPI) - Baseline | Baseline Visit
  The Denture Plaque Index (DPI) is scored by removing the denture, placing it in a bath of disclosing solution for 30 seconds, rinsing it under lukewarm water for 15 seconds, and assigning a score to each of four quadrants (upper and lower, and lingual and buccal) as follows: 0=no plaque, 1=light plaque (1-25% of area covered), 2=moderate plaque (26-50% of area covered), 3=heavy plaque (51-75% of area covered), or 4=very heavy plaque (76 100% of area covered). DPI is reported as the mean score of all quadrants and lower scores are better.
Aim2 - Denture Plaque Index Score (DPI) - 4 Months | 4 Months Follow-up Visit
  The Denture Plaque Index (DPI) is scored by removing the denture, placing it in a bath of disclosing solution for 30 seconds, rinsing it under lukewarm water for 15 seconds, and assigning a score to each of four quadrants (upper and lower, and lingual and buccal) as follows: 0=no plaque, 1=light plaque (1-25% of area covered), 2=moderate plaque (26-50% of area covered), 3=heavy plaque (51-75% of area covered), or 4=very heavy plaque (76 100% of area covered). DPI is reported as the mean score of all quadrants and lower scores are better.
Aim2 - Change in Denture Plaque Index Score (DPI) - 4 Months | Change from Baseline to 4 months
  The Denture Plaque Index (DPI) is scored by removing the denture, placing it in a bath of disclosing solution for 30 seconds, rinsing it under lukewarm water for 15 seconds, and assigning a score to each of four quadrants (upper and lower, and lingual and buccal) as follows: 0=no plaque, 1=light plaque (1-25% of area covered), 2=moderate plaque (26-50% of area covered), 3=heavy plaque (51-75% of area covered), or 4=very heavy plaque (76 100% of area covered). DPI is reported as the mean score of all quadrants and lower scores are better.
Aim3 - Plaque Index Score for Long-Term Care (PI-LTC) - Baseline | Baseline Visit
  The Plaque Index for Long-Term Care (PI-LTC) is a modification of the Simplified Oral Hygiene Index. It is derived by separately scoring the buccal and lingual surfaces of six sextants in the mouth (left, front, and right regions of the upper and lower jaw), resulting in 12 separate observations for residents with a full set of teeth; sextants not containing teeth do not receive a score. Within each sextant, the tooth surface with the worst plaque is scratched using an explorer and assigned a score (0=no plaque or stain present; 1=soft plaque covering not more than one third of the tooth surface or presence of extrinsic stains without other plaque regardless of surface area covered; 2=soft plaque covering between one third and two thirds of the tooth surface; or 3=soft plaque covering more than two thirds of the exposed tooth surface). PI-LTC scores range from 0-3 and are the average sextant score. Lower scores are better.
Aim3 - Plaque Index Score for Long-Term Care (PI-LTC) - 4 Months | 4 Months Follow-up Visit
  The Plaque Index for Long-Term Care (PI-LTC) is a modification of the Simplified Oral Hygiene Index. It is derived by separately scoring the buccal and lingual surfaces of six sextants in the mouth (left, front, and right regions of the upper and lower jaw), resulting in 12 separate observations for residents with a full set of teeth; sextants not containing teeth do not receive a score. Within each sextant, the tooth surface with the worst plaque is scratched using an explorer and assigned a score (0=no plaque or stain present; 1=soft plaque covering not more than one third of the tooth surface or presence of extrinsic stains without other plaque regardless of surface area covered; 2=soft plaque covering between one third and two thirds of the tooth surface; or 3=soft plaque covering more than two thirds of the exposed tooth surface). PI-LTC scores range from 0-3 and are the average sextant score. Lower scores are better.
Aim3 - Change in Plaque Index Score for Long-Term Care (PI-LTC) - 4 Months | Change from Baseline to 4 months
  The Plaque Index for Long-Term Care (PI-LTC) is a modification of the Simplified Oral Hygiene Index. It is derived by separately scoring the buccal and lingual surfaces of six sextants in the mouth (left, front, and right regions of the upper and lower jaw), resulting in 12 separate observations for residents with a full set of teeth; sextants not containing teeth do not receive a score. Within each sextant, the tooth surface with the worst plaque is scratched using an explorer and assigned a score (0=no plaque or stain present; 1=soft plaque covering not more than one third of the tooth surface or presence of extrinsic stains without other plaque regardless of surface area covered; 2=soft plaque covering between one third and two thirds of the tooth surface; or 3=soft plaque covering more than two thirds of the exposed tooth surface). PI-LTC scores range from 0-3 and are the average sextant score. Lower scores are better.
Aim3 - Gingival Index Score for Long-Term Care (GI-LTC) - Baseline | Baseline Visit
  The Gingival Index for Long-Term Care (GI-LTC) is a modification of the Gingival Index. Within each sextant, the most inflamed gingival surface is identified, swept using an explorer, and assigned a score (0=no inflammation; 1=mild inflammation, slight change in color, little change in texture; 2=moderate inflammation, glazing, redness, edema, and/or hypertrophy; or 3=severe inflammation, marked redness, edema and/or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration). Overall GI-LTC scores range from 0-3 and are the average sextant score. Buccal and lingual surfaces scores also are calculated. Lower scores are better.
Aim3 - Gingival Index Score for Long-Term Care (GI-LTC) - 4 Months | 4 Months Follow-up Visit
  The Gingival Index for Long-Term Care (GI-LTC) is a modification of the Gingival Index. Within each sextant, the most inflamed gingival surface is identified, swept using an explorer, and assigned a score (0=no inflammation; 1=mild inflammation, slight change in color, little change in texture; 2=moderate inflammation, glazing, redness, edema, and/or hypertrophy; or 3=severe inflammation, marked redness, edema and/or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration). Overall GI-LTC scores range from 0-3 and are the average sextant score. Buccal and lingual surfaces scores also are calculated. Lower scores are better.
Aim3 - Change in Gingival Index Score for Long-Term Care (GI-LTC) - 4 Months | Change from Baseline to 4 months
  The Gingival Index for Long-Term Care (GI-LTC) is a modification of the Gingival Index. Within each sextant, the most inflamed gingival surface is identified, swept using an explorer, and assigned a score (0=no inflammation; 1=mild inflammation, slight change in color, little change in texture; 2=moderate inflammation, glazing, redness, edema, and/or hypertrophy; or 3=severe inflammation, marked redness, edema and/or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration). Overall GI-LTC scores range from 0-3 and are the average sextant score. Buccal and lingual surfaces scores also are calculated. Lower scores are better.
Aim3 - Denture Plaque Index Score (DPI) - Baseline | Baseline Visit
  The Denture Plaque Index (DPI) is scored by removing the denture, placing it in a bath of disclosing solution for 30 seconds, rinsing it under lukewarm water for 15 seconds, and assigning a score to each of four quadrants (upper and lower, and lingual and buccal) as follows: 0=no plaque, 1=light plaque (1-25% of area covered), 2=moderate plaque (26-50% of area covered), 3=heavy plaque (51-75% of area covered), or 4=very heavy plaque (76 100% of area covered). DPI is reported as the mean score of all quadrants and lower scores are better.
Aim3 - Denture Plaque Index Score (DPI) - 4 Months | 4 Months Follow-up visit
  The Denture Plaque Index (DPI) is scored by removing the denture, placing it in a bath of disclosing solution for 30 seconds, rinsing it under lukewarm water for 15 seconds, and assigning a score to each of four quadrants (upper and lower, and lingual and buccal) as follows: 0=no plaque, 1=light plaque (1-25% of area covered), 2=moderate plaque (26-50% of area covered), 3=heavy plaque (51-75% of area covered), or 4=very heavy plaque (76 100% of area covered). DPI is reported as the mean score of all quadrants and lower scores are better.
Aim3 - Change in Denture Plaque Index Score (DPI) - 4 Months | Change from Baseline to 4 months
  The Denture Plaque Index (DPI) is scored by removing the denture, placing it in a bath of disclosing solution for 30 seconds, rinsing it under lukewarm water for 15 seconds, and assigning a score to each of four quadrants (upper and lower, and lingual and buccal) as follows: 0=no plaque, 1=light plaque (1-25% of area covered), 2=moderate plaque (26-50% of area covered), 3=heavy plaque (51-75% of area covered), or 4=very heavy plaque (76 100% of area covered). DPI is reported as the mean score of all quadrants and lower scores are better.

SECONDARY OUTCOMES:
Aim2 - Cumulative incidence of pneumonia | Cumulative from Baseline to Completion (up to 8 months)
  The total number of diagnosed cases of pneumonia
Aim2 - Cumulative incidence of hospitalizations | Cumulative from Baseline to Completion (up to 8 months)
  The total number of hospitalizations
Aim3 - Cumulative incidence of pneumonia | Cumulative from Baseline to Completion (up to 4 months)
  The total number of diagnosed cases of pneumonia
Aim3 - Cumulative incidence of hospitalizations | Cumulative from Baseline to Completion (up to 4 months)
  The total number of hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: Sheryl Zimmerman, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be shared after deidentification.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Deidentified individual data that supports the results will be shared beginning 3 months and ending 5 years following article publication.
Access Criteria: An investigator who proposes to use the data must have approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and execute a data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Cao Y, Liu C, Lin J, Ng L, Needleman I, Walsh T, Li C. Oral care measures for preventing nursing home-acquired pneumonia. Cochrane Database Syst Rev. 2022 Nov 16;11(11):CD012416. doi: 10.1002/14651858.CD012416.pub3. PMID 36383760

DOCUMENTS (1):
  • Informed Consent Form (2024-06-28): https://cdn.clinicaltrials.gov/large-docs/00/NCT03892200/ICF_000.pdf